CLINICAL TRIAL: NCT03596671
Title: A Prospective Study to Assess the Efficacy and Safety of the BlueWind RENOVA iStim™ System in the Treatment of Patients Diagnosed With Overactive Bladder (OASIS - OverActive Bladder StImulation System Study)
Brief Title: BlueWind RENOVA iStim™ System for the Treatment of OAB
Acronym: OASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BlueWind Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G02-CLP-0002
Record Dates: First submitted 2018-07-01; First posted 2018-07-24 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Treatment of Patients Suffering From Overactive Bladder (OAB)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment arm (Experimental): RENOVA iStim™ System implanted patients
  Interventions: Device: RENOVA iStim™ System

INTERVENTIONS:
Device: RENOVA iStim™ System — Tibial implantable neuromodulation device

SUMMARY:
The OASIS study is prospective, interventional, multi-center study to evaluate the safety and efficacy of the BlueWind RENOVA iStim™ implantable tibial neuromodulation System for the treatment of patients diagnosed with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 or greater (21 in the US)
* More than or equal to 6 months history of UUI diagnosis
* Patient who is mentally competent with the ability to understand and comply with the requirements of the study

Exclusion Criteria:

* Any significant medical condition that is likely to interfere with study procedures
* Patients who are breastfeeding
* Predominant stress incontinence
* Have a life expectancy of less than 1 year
* Diagnosis of interstitial cystitis or bladder pain syndrome as defined by either American Urological Association (AUA) or European Association of Urology (EAU) guidelines

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2025-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Heesakkers, MD, Principal Investigator — Maastricht University Medical Centre
Locations (23):
- United States (14):
  - University of California Irvine, Orange, California
  - Kaiser Permanente, San Diego, California
  - Norwalk Urology, Norwalk, Connecticut
  - Florida Urology Partners, Tampa, Florida
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology - Hanover, Hanover, Maryland
  - Chesapeake Urology - Owing Mills, Owings Mills, Maryland
  - Minnesota Urology, Woodbury, Minnesota
  - Adult Pediatric Urology & Urogynecology, Omaha, Nebraska
  - Duke Urogynecology, Durham, North Carolina
  - Southern Urogynocology, West Columbia, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - University of Washington, Seattle, Washington
- Belgium (2):
  - University Hospital Antwerp, Antwerp
  - UZ Leuven, Leuven
- Netherlands (5):
  - Rijnstate Hospital, Arnhem
  - Academic Hospital Maastricht, Maastricht
  - Radboud University Medical Center, Nijmegen
  - UMC Utrecht, Utrecht
  - Isala, Zwolle
- United Kingdom (2):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - Imperial College, St. Mary's Hospital, London

REFERENCES:
- [Derived] Heesakkers JPFA, Toozs-Hobson P, Sutherland SE, Digesu A, Amundsen CL, McCrery RJ, De Wachter S, Kean ER, Martens F, Benson K, Ferrante KL, Cline KJ, Padron OF, Giusto L, Lane FL, Witte LPW, Dmochowski RR. Two-Year Efficacy and Safety Outcomes of the Pivotal OASIS Study Using the Revi System for Treatment of Urgency Urinary Incontinence. J Urol. 2025 Mar;213(3):323-332. doi: 10.1097/JU.0000000000004328. Epub 2024 Nov 25. PMID 39585851

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started (Screened for Eligibility) | 282
Implanted | 151
6 Months Follow-up | 144
Completed (12 months follow-up) | 140
Not Completed | 142

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Captured for US participants only.
  Participants
    Race: Black or African American | 3
    Race: White | 83
    Race: Other | 1
    Race: Not Collected - European Participants | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Captured for US participants only.
  Participants
    Ethnicity: Hispanic or Latino | 6
    Ethnicity: Not Hispanic or Latino | 81
    Ethnicity: Not Collected - European Participants | 64
Region of Enrollment [Number; unit: participants]
  Netherlands | 25
  Belgium | 11
  United States | 87
  United Kingdom | 28
Height [Mean (Standard Deviation); unit: cm] | 165.4 (6.6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.2 (6.9)
Time since OAB diagnosis [Count of Participants; unit: Participants] — Population: Duration unreported in 1 participant
  Participants
    number analyzed (Participants) | 150
    < 6 months | 2
    6 months to 1 year | 7
    1-5 years | 44
    > 5 years | 97

OUTCOME MEASURES:

1. Primary Outcome: ≥50% Decrease in Mean Urinary Urgency Incontinence (UUI) Episodes
Description: Proportion of responders at 6 months post system activation as demonstrated by ≥50% improvement in average number of urgency related incontinence episodes, measured by 7-day Patient Voiding Diary.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of Responders
Arm/Group | Treatment Arm
Number analyzed (Participants) | 151
Percentage of Responders | 76.4 [68.7 to 82.6]

2. Primary Outcome: Safety - Number of Participants With Adverse Events
Description: The primary safety endpoint was to assess adverse events from implantation to 12-months post-activation (Treatment Emergent Adverse Events).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 151
Participants
  Subjects with reported Adverse Events (AEs) | 117
  Subjects with procedure-related AEs (CEC adjudicated) | 16
  Subjects with device-related AEs (CEC adjudicated) | 6
  Subjects with wound-related AEs (CEC adjudicated) | 10
  Subjects with a reported Serious Adverse Event (SAE) (CEC Adjudicated) | 13

ADVERSE EVENTS:
Time Frame: 12 months
Description: Safety events have been reported for all subjects in which an implant of the BlueWind device was attempted. All subjects in whom an implant was attempted were successfully implanted.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/151
Serious Adverse Events (participants affected / at risk) | 13/151
Other Adverse Events (participants affected / at risk) | 34/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=151)
COVID-19 (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Herpes zoster meningitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Post - traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=151)
Urinary Tract Infection (Infections and infestations) | 34 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03596671/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03596671/SAP_001.pdf